CLINICAL TRIAL: NCT07079150
Title: Real-world Study Evaluating the Long-term Outcomes of Pegylated Interferon α-2b Treatment in the Families With Clusters of HBV Infection and Unfavorable Prognosis - A Prospective, Controlled, Multicenter, Cohort Study
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2024LSYY-468
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Hepatitis B, Chronic (CHB); Hepatitis B; Hepatitis B Virus (HBV)
Keywords: hepatitis B; family cluster; interferon; antiviral therapy; cirrhosis; hepatocellular carcinoma
MeSH Terms: conditions — Hepatitis B; Bronchiolitis Obliterans Syndrome; Fibrosis; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Peg IFN-α-2b combined with NAs therapy for non-cirrhotic group
  Interventions: Drug: Peg IFN-α-2b
- NAs monotherapy for non-cirrhotic group
- Peg IFN-α-2b combined with NAs therapy for cirrhotic group
  Interventions: Drug: Peg IFN-α-2b
- NAs monotherapy for cirrhotic group

INTERVENTIONS:
Drug: Peg IFN-α-2b — In the treatment of Peg IFNα-2b combined with NAs (Peg IFN combined treatment group), the treatment of Peg IFNα-2b should be no less than 48 weeks. The initial therapeutic dose of Peg IFNα-2b and the subsequent adjusted dose will be individualized determined by clinicians based on the specific condition of the patients. In the NAs monotherapy group, entecavir (ETV), tenofovir fumarate disoproxil (TDF), tenofovir propofol fumarate (TAF), and emitenofovir (TMF) were used for treatment for no less than 48 weeks, and Peg IFN was not added or switched for treatment.
  Groups: Peg IFN-α-2b combined with NAs therapy for cirrhotic group; Peg IFN-α-2b combined with NAs therapy for non-cirrhotic group

SUMMARY:
Chronic hepatitis B can develop into cirrhosis and liver cancer, which seriously endangers the life and health of people. In China, HBV is mainly transmitted from mother to child, showing the phenomenon of family clusters. Similarly, cirrhosis and hepatocellular carcinoma occur in familial clusters. Familial clusters of HBV infection with unfavorable prognoses refers to HBV-infected patients from two consecutive generations of blood relatives, with at least one family member diagnosed with hepatitis B-related cirrhosis or hepatocellular carcinoma (HCC). Previous family investigations have shown that the risk and harm of HBV-related cirrhosis and hepatocellular carcinoma are significantly higher in families with familial clusters of HBV infection with unfavorable prognoses than in the general population.

Currently, antiviral drugs used for CHB mainly include nucleoside analogues (NAs) and interferon-alpha (mainly pegylated interferon-alpha, Peg IFN). NAs mainly inhibits viral replication by blocking the reverse transcription process, but it cannot effectively inhibit the expression of viral proteins such as HBsAg, and rarely achieves clinical cure. Multiple clinical studies have shown that the use of NAs reduces the incidence of cirrhosis decompensation, HCC, and death in patients with CHB compared to untreated or placebo-treated patients. Despite long-term treatment with first-line NAs drugs, CHB patients continue to be at risk of developing hepatocellular carcinoma. Peg IFN α-2b injection is the first-line drug of choice for antiviral treatment of chronic hepatitis B, and its main mechanism of action includes anti-HBV, anti-fibrosis, anti-tumor and regulation of immune response. In 2024, a randomized controlled multicenter study showed that Peg IFN α-2b combined with NAs therapy could effectively prevent hepatocellular carcinoma in CHB patients. There is sufficient evidence in clinical practice that long-term antiviral therapy, whether NAs or Peg IFN α-2b, reduces the risk of cirrhosis, hepatocellular carcinoma, and death in patients with CHB. In conclusion, early antiviral therapy can reduce the risk of developing hepatitis B cirrhosis and hepatocellular carcinoma in CHB patients with familial clusters of HBV infection with unfavorable prognoses.

The goal of this observational study is to explore the evaluation of pegylated interferon α-2b combined with first-line NAs on the long-term outcome of CHB antiviral therapy with cirrhosis and HCC progression as the main observation targets, compared with only use of NAs in the context of familial clusters of HBV infection with unfavorable prognoses. It is intended to provide high-quality evidence-based medical evidence for the treatment and follow-up of CHB, explore optimal clinical decision-making, and provide global clinical data for the improvement and evaluation of this difficult-to-treat population. The main question it aims to answer is: Can Peg IFN-α-2B combined with NAs therapy improve the long-term outcomes of this particular population of familial clusters of HBV infection with unfavorable prognoses compared to first-line NAs monotherapy? Patients with familial clusters of HBV infection with unfavorable prognoses using Peg IFN-α-2B combined with NAs therapy and NAs monotherapy will be collected laboratory and medical examination data at specified follow-up points, and recorded adverse events and drug combinations in detail for 7 years.

DETAILED DESCRIPTION:
Study Backgrounds: Chronic hepatitis B (CHB) refers to an infectious disease characterized primarily by liver lesions that persist for more than six months, caused by the hepatitis B virus (HBV). According to the World Health Organization, in 2019, the global prevalence of HBsAg in the general population was 3.8%, with approximately 296 million chronic HBV infections, 1.5 million new HBV infections, and 820,000 deaths due to liver failure, cirrhosis, or hepatocellular carcinoma (HCC) related to HBV infection. Data released by the Polaris International Epidemiology Collaboration in December 2023 on the progress of eliminating hepatitis B in China showed that there are 79.742 million chronic HBV infections in China, with a diagnosis rate of only 24% and an annual treatment rate of only 15%, with more than 450,000 annual deaths related to hepatitis B. According to the National Disease Prevention and Control Bureau's report on nationally notifiable infectious diseases, there are about 1 million new cases of hepatitis B in China each year, with 1.05 million new cases in 2023, making it the fourth leading cause of death from infectious diseases in China.

HBV can trigger host antiviral immunity through direct and indirect mechanisms, leading to liver inflammation, fibrosis, and cirrhosis. Additionally, HBV DNA can integrate into the host genome, activating oncogenes, causing chromosomal instability, and epigenetic changes, ultimately leading to HCC. The risk factors for the development of cirrhosis mainly include host factors (older age, male, HBeAg seroconversion at >40 years old, persistently elevated ALT), viral factors (HBV DNA > 2,000 IU/mL, persistently positive HBeAg, C genotype), co-infections (HCV, HDV, HIV), and other liver damage factors (such as alcohol consumption or obesity). Without antiviral treatment, the annual incidence of cirrhosis in CHB patients is 2-10%. The annual incidence of decompensated cirrhosis progressing from compensated cirrhosis is 3-5%, with a 5-year survival rate of 14-35%. The annual incidence of HCC in non-cirrhotic HBV-infected individuals is 0.2-1.0%, while in cirrhotic patients, it is 3-6%. Factors such as age >40, male, cirrhosis, family history of HCC, high-level replication of HBV, alcohol consumption, smoking, coexisting diabetes, obesity, and exposure to aflatoxins are all associated with a high incidence of HCC. In China, chronic HBV infection is the main cause of HCC, accounting for about 86% of HCC occurrences. As the fourth most common malignant tumor and the second leading cause of cancer-related deaths in China, HCC poses a serious threat to the lives and health of people. CHB and HBV-related diseases such as cirrhosis and HCC impose a huge disease burden on China, significantly affecting families and representing one of China's major public health challenges.

According to the Guidelines for the Prevention and Treatment of Chronic Hepatitis B (2022 Edition), the main goal of CHB treatment is to maximize long-term suppression of HBV replication, alleviate hepatocyte inflammation and necrosis, and liver fibrosis, thereby delaying and reducing the occurrence of liver failure, decompensated cirrhosis, HCC, and other complications. The current clinically used antiviral drugs for CHB mainly include nucleoside (tide) analogs (NAs) and interferon-α (IFN-α) (currently pegylated interferon-α). Antiviral therapy can slow the progression of CHB to cirrhosis and HCC. NAs mainly inhibit viral replication by blocking the reverse transcription process and are all oral medications, which are convenient to use and well-tolerated. However, since they cannot directly inhibit the transcriptional activity of cccDNA, they cannot effectively suppress the expression of viral proteins such as HBsAg, rarely achieving clinical cure. HBsAg decreases slowly during treatment, with an average annual seroconversion rate of 0-1.3% under long-term treatment, thus requiring long-term medication maintenance. Moreover, despite long-term NAs therapy with first-line drugs, there is still a stable and continuous risk of HCC over time, with an increasing annual incidence. Pegylated interferon α-2b (Peg IFN α-2b) is a first-line drug for the antiviral treatment of chronic hepatitis B, with main effects including anti-HBV, anti-fibrotic, antitumor, and immune regulation mechanisms. IFN-α exerts dual effects by enhancing host immune responses and direct antiviral actions at multiple levels. In addition to inhibiting the viral replication process, it affects the transcriptional inhibition of cccDNA, the degradation of cccDNA, and the clearance of HBV-infected cells, inducing a sustained immune response, which is more conducive to virus clearance. During treatment, HBsAg decreases more rapidly in some patients, with previous studies observing an HBsAg seroconversion rate of 2.8-7% at 48 weeks of IFN-α monotherapy, higher than that of NA monotherapy, and continued benefits after discontinuation of IFN-α. Therefore, IFN-α can promote the reduction of incidence and mortality related to liver cirrhosis and HCC. Additionally, IFN-α can inhibit tumor angiogenesis and tumor cell proliferation, which can explain its role in preventing the recurrence of HCC after surgery for HBV-related HCC and in preventing the occurrence of HCC in CHB patients. However, IFN-α preparations require subcutaneous injection and are relatively common in adverse reactions such as bone marrow suppression and flu-like symptoms, with relatively poor tolerance. The Guidelines for the Prevention and Treatment of Chronic Hepatitis B (2022 Edition) indicate that for eligible patients with CHB treated with NAs, the combination of Peg-IFN-α can lead to functional cure in some patients. Although antiviral treatment against HBV can significantly reduce the risk of liver cancer, it cannot completely avoid the occurrence of HCC. Current research on the advantages and disadvantages of different antiviral treatment regimens for CHB, especially the long-term prognosis differences in the incidence of decompensated cirrhosis and HCC after different antiviral treatment regimens, is insufficient.

HBV is mainly transmitted through mother-to-child, blood, and sexual contact, with mother-to-child transmission being the most common. In China, HBV infection is mainly through mother-to-child transmission, showing a family clustering phenomenon. In addition, the occurrence of cirrhosis and hepatocellular carcinoma also has a family clustering nature. Although free hepatitis B vaccination is implemented in various parts of China, due to unbalanced regional economic development, different levels of social education and culture, and uneven individual health knowledge, HBV infection cannot be completely blocked, leading to a significant family clustering of HBV infection, showing a trend of younger-age and high incidence. Many studies and guidelines have pointed out that a family history of HBV-related cirrhosis or HCC is an independent risk factor for the progression of liver disease and the occurrence of HCC. In a large cohort study of CHB patients, the odds ratio (OR) for HCC occurrence in non-cirrhotic patients with a family history of liver cancer was 32.9 times. A survey study of 102 family lineages at the First Affiliated Hospital of Xi'an Jiaotong University in China showed that the prevalence rates of cirrhosis among probands, first-degree relatives (siblings, parents, and children of the proband), second-degree relatives (siblings, parents, and children of the first-degree relatives), and non-relatives were 57.4%, 29.2%, 11.9%, and 8.7%, respectively. The prevalence rates of HCC were 28.7%, 21.8%, 1.4%, and 4.3%, respectively. The average ages at which cirrhosis was diagnosed in probands, first-degree relatives, and second-degree relatives were 57±9.91, 47±9.96, and 38±10.35 years, respectively. The average ages at which HCC was diagnosed were 60±7.92, 49±8.57, and 41±3.35 years, respectively. As the degree of kinship becomes more distant, the rate of HBV infection decreases, but the age of onset advances, the prevalence rates of cirrhosis and HCC decrease, and the prevalence rates of cirrhosis and HCC among different degrees of relatives in families with adverse outcomes of HBV infection are significantly higher than in the general population. Therefore, the risks and harms of HBV-related cirrhosis and HCC in families with unfavorable prognoses of HBV infection are significantly higher than in the general population.

Clinical practice has ample evidence showing that long-term antiviral treatment, whether with NAs or IFN-α, can reduce the risk of HCC in patients with chronic hepatitis B. The "Consensus on Secondary Prevention of Primary Liver Cancer (2021 Edition)" has indicated that the prevention of HCC in populations with chronic HBV/HCV infection and other chronic liver diseases is secondary prevention, and antiviral treatment for HBV is treatment to control the cause. Previous studies have shown that treatment based on PEG-IFN-α can further reduce the risk of liver cancer by more than 85% on the basis of NAs. Therefore, if antiviral treatment can be used as early as possible to achieve HBsAg seroconversion or serum conversion in patients with adverse outcomes of family clustering of HBV, it will reduce the risk of patients developing hepatitis B cirrhosis and HCC. Currently, there is insufficient research on the long-term prognosis differences in the incidence of decompensated cirrhosis and HCC after different antiviral treatment regimens in patients with CHB from families with unfavorable prognoses of HBV infection. There is an urgent clinical need for high-quality clinical studies with large samples and long-term follow-up to provide evidence-based support for the optimization of antiviral regimens.

This study aims to establish a prospective, controlled, multicenter, observational cohort study design to explore, in the context of families with unfavorable prognoses of family clustering of HBV infection, the impact of Peg IFN α-2b combined with NAs on the long-term outcomes of antiviral treatment for CHB, with cirrhosis and HCC progression as the main observation targets, compared with monotherapy with first-line NAs: referring to the use of entecavir (ETV), tenofovir disoproxil fumarate (TDF), tenofovir alafenamide fumarate (TAF), or tenofovir amibufenamide (TMF). The study intends to provide high-quality evidence-based medical evidence for the treatment and follow-up of CHB, explore the best clinical decisions, and provide globally promotable clinical data for the improvement and evaluation of this difficult-to-treat population.

The study plans to enroll patients from multiple research centers across the country, collecting data on antiviral (Peg IFN or NAs) treatments from CHB patients with a family history of unfavorable prognoses associated with HBV infection, and conducting a prospective real-world study. Standard methods are used in the study to collect data, conduct analysis, and evaluation. In this study, patients in each group choose different treatment plans based on the judgment of the clinician and the wishes of the patient. The treatment plans included in the study observation are combination therapy with Peg IFN α-2b and NAs (Peg IFN combination therapy group), and monotherapy with NAs (nucleos(t)ide monotherapy group), where interferon treatment is no less than 48 weeks. The initial therapeutic dose of Peg IFN α-2b and subsequent dose adjustment will be determined individually by the clinician based on the patient's specific condition. NAs include ETV, TDF, TAF, or TMF. During the study, if patients experience virological breakthrough, they may add or switch to other NAs treatments. This study does not conduct any interventions, only observes and records the treatment situation, collects data from laboratory tests, medical examinations, and other data at specified follow-up points, and records adverse events and concomitant medications in detail. During the treatment process of the two groups of patients, it is allowed to change the type of nucleos(t)ide medication according to the patient's condition or wishes, and detailed records must be kept.

Since this study is non-interventional, to ensure a higher follow-up rate among patients, we will strengthen education and reminders during the initial and follow-up visits, informing patients of the next scheduled follow-up appointment. The database software system will have a feature that regularly prompts the principal investigators at each center about the recommended follow-up time points, reminding the center's physicians to follow up with patients and collect and enter data as needed. Additionally, we will distribute patient education manuals that include follow-up record forms, encouraging patients to adhere to regular follow-ups and to regularly record their own follow-up examination results, thereby understanding their condition and treatment effects.

Before considering a patient as "lost to follow-up," trained research personnel at each center will make every effort to contact the patient and keep them on the registration list. If no response is obtained from the patient, we will contact the patient's designated relatives to confirm whether the reason for the patient's non-response is health-related and to ascertain the patient's status. If the patient has died, we will determine the time and cause of death.

During the follow-up period, efforts should be made to comprehensively collect information on adverse reactions in patients undergoing antiviral treatment, including patient conditions, reporter conditions, suspected and concomitant medications, and the occurrence of adverse reactions. If it is difficult to obtain comprehensive information, the four essential elements of information should be obtained first (identifiable patient, identifiable reporter, suspected medication, adverse reaction). For various channels through which adverse reaction information is received during patient follow-up, there should be original records. Records should be true, accurate, objective, and properly preserved. Original records can be paper records, electronic documents, audio recordings, or website screenshots, etc. Routine collection methods such as telephone records and doctor's visits should have original record forms. All original records should clearly indicate the date on which the adverse reaction to the medication was obtained and the name and contact information of the first receiver.

Each subject will be assigned a screening number, which is a 6-digit number composed of a center number and an enrollment sequence number, with the first 3 digits being the center number and the last 4 digits being the screening sequence number. For example, the 7th subject at the 3rd center, their screening number would be 00300007. Once a subject is numbered, that number will not be reused.

Relevant materials for this study will be obtained after the patient signs the informed consent form, through direct access via disease registration systems, electronic medical records, or based on reliable medical history provided by the patient and presented examination reports.

Data entry and modification of paper case report forms are the responsibility of trained researchers at each center and are stored in a dedicated, fixed filing cabinet, which is locked with a key kept by a designated person at each research center.

During the study, the subject's case report forms will also be stored in electronic format. The electronic case report form is designed and constructed by the data manager based on the study protocol and the original case report form.

Data will be extracted in an unstructured format. Unstructured data refers to medical data recorded verbatim, including textual descriptions and visual descriptions of medical information, such as medical records, images of doctor's notes, or narrative fields in databases. Researchers or clinical research coordinators (CRC) fill out the case report forms to manually extract unstructured data into a set of predefined data tables, which are then input into the electronic case report form (eCRF) through a standardized electronic case report form interface.

The eCRFs for this study are stored in a database. The study uses data storage software to establish the database, which is maintained and quality-controlled by trained members of the study group, without the involvement of third parties. Data entry and modification are the responsibility of trained researchers at each center, and the data should be sourced from original record forms and laboratory test reports and should be consistent with the original documents. Any observations or examination results in the study should be recorded in tables or databases in a timely, accurate, complete, clear, standardized, and truthful manner. The data manager, a member of the study group, is responsible for reviewing and managing the entered data. In case of any questions about the data, the data manager will send queries to the researchers at each center who entered the data. Researchers who entered the data should promptly respond to the queries sent by the data manager, and the data manager may send further queries if necessary.

The entry and modification of paper CRF data in this study are the responsibility of trained researchers at each center and are stored in a dedicated, fixed filing cabinet, which is locked with a key kept by a designated person at each research center.

This study is a real-world prospective controlled study that does not involve statistical hypothesis testing or sample size estimation. The study will be conducted across multiple centers, planning to include 1200 non-cirrhosis and 300 compensated cirrhosis patients who meet the inclusion criteria and do not meet the exclusion criteria. In the non-cirrhotic cohort, the Peg IFN combination therapy group plans to enroll 600 patients, and the nucleos(t)ide group plans to enroll 600 patients; in the compensated cirrhosis cohort, the Peg IFN combination therapy group plans to enroll 150 patients, and the nucleos(t)ide monotherapy group plans to enroll 150 patients.

The principal investigator will organize data management and implement research project training to ensure that the study is conducted in a standardized and reasonable manner, with the completion of case report forms or study records following GCP principles and the study protocol. All data and materials can be audited; to ensure the reliability of the study data, all observations and findings must be verifiable. Quality control will be applied at every stage of the study to ensure the reliability of all data and the accuracy of research procedures. The principal investigator will ensure that researchers adhere to the study protocol, confirm the accuracy of the data and the completeness of the records and reports, and ensure that informed consent is obtained from all subjects before the study begins. Any deviations from or violations of the protocol will be reported to the ethics committee in a timely manner.

The research team will establish the following standard operating procedures in data management, implementing quality control procedures at every stage of research implementation and data processing to ensure the standardization and reliability of research implementation and data operations.

Statistical analysis:

Analysis Sets:

Full Analysis Set (FAS): In accordance with the principles of Intention-to-Treat (ITT), includes all enrolled subjects.

Per-Protocol Set (PPS): Within the FAS population, the PPS includes all subjects who have completed the treatment as specified in the protocol and have not seriously violated the trial protocol. Efficacy analysis will use both FAS and PPS.

Safety Analysis Set (SS): Includes all subjects who have been enrolled and have used the study medication at least once.

The determination of all analysis sets will be made at the data review meeting. Statistical analysis software will use SAS V9.4 or higher or R statistical analysis software.

Descriptive statistics for quantitative indicators will calculate the number of cases, mean, standard deviation, median, minimum value, and maximum value. For qualitative indicators, the number of cases and percentages will be described, with the calculation of percentages based on non-missing data as the denominator, unless otherwise specified, using chi-square tests or Fisher's exact probability method for inter-group rate comparisons. For survival data, the Kaplan-Meier method will be used to estimate the median time and its 95% confidence interval (CI), and the log-rank test will be used for inter-group comparisons.

All statistical tests will use two-sided tests, and a P-value less than 0.05 will be considered statistically significant for the differences tested (unless otherwise specified). For more details, see the attached statistical analysis plan.

The Intention-to-Treat population will be used for the analysis of baseline data. Subject characteristics include demographic data, baseline medical history, and disease characteristics, etc. According to the numerical characteristics of the variables, the age, height, weight, and other quantitative data of the two groups of subjects will be compared using analysis of variance and/or Kruskal-Wallis rank sum tests; qualitative variables such as gender, ethnicity, drug allergy history, smoking and drinking history, drug abuse, family history, allergy history, hepatitis B infection history, hepatitis B treatment history, and past comorbidity history of the two groups of subjects will be compared using chi-square tests and/or Fisher's exact probability method.

Primary Efficacy Endpoint Analysis:

1. In the non-cirrhosis population of chronic HBV-infected patients from families with unfavorable prognoses familial clustering of HBV infection, the number and percentage of cirrhosis and HCC cases at 240 weeks (5 years) and 336 weeks (7 years) of treatment for both the nucleos(t)ide group and the Peg IFN combination therapy group will be statistically analyzed. The incidence rates and 95% CI for each group will be calculated, and inter-group rate comparisons will be made using chi-square tests or Fisher's exact probability method.
2. In the compensated cirrhosis population of chronic HBV-infected patients from families with unfavorable prognoses familial clustering of HBV infection, the number and percentage of decompensated cirrhosis and HCC cases at 240 weeks (5 years) and 336 weeks (7 years) of treatment for both the nucleos(t)ide group and the Peg IFN combination therapy group will be statistically analyzed. The incidence rates and 95% CI for each group will be calculated, and inter-group rate comparisons will be made using chi-square tests or Fisher's exact probability method.

Secondary Efficacy Endpoint Analysis:

1. In the sub-populations, the overall survival time (OS) for patients in each treatment group will be described statistically. The median OS (mOS) and its 95% CI will be estimated using the Kaplan-Meier method, and survival curves will be plotted. Inter-group comparisons will be made using the log-rank test.
2. In the sub-populations, the time to the occurrence of cirrhosis and liver cancer for patients in each treatment group will be described statistically. The median time to occurrence and its 95% CI will be estimated using the Kaplan-Meier method, and survival curves will be plotted. Inter-group comparisons will be made using the log-rank test.
3. In the sub-populations, the number and percentage of patients with HBsAg seroconversion and HBeAg seroconversion (for those who are HBeAg-positive) will be described statistically every 24 weeks for both treatment groups.
4. In the sub-populations, the levels of HBV DNA, HBsAg, and HBeAg will be described statistically every 24 weeks for both treatment groups.

Safety Analysis:

Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). Adverse events will be assessed and graded according to the NCI CTCAE version 5.0.

Descriptive statistics will be conducted for the occurrence of various adverse events (such as the number of subjects experiencing the event, percentage, and frequency of adverse event occurrences), and all adverse events, adverse events related to the study medication, adverse events of grade 3 or higher, and serious adverse events will be summarized according to the System Organ Class (SOC) and Preferred Term (PT).

For other safety indicators, including physical examinations, vital signs, clinical laboratory tests, imaging examinations, concomitant medications, etc., descriptive statistics will be conducted, and any abnormal changes in the examination results will be summarized.

Ethical Considerations:

The Ethics Committee of the First Affiliated Hospital of Xi'an Jiaotong University is responsible for reviewing the scientific and ethical rationality of the trial protocol. The Ethics Committees of each participating institution, under the premise of accepting the review opinions of the leading unit's Ethics Committee, are responsible for reviewing the feasibility of the trial at their institution. At the same time, for all selected patients, informed consent will be signed. If a patient decides to participate in this study, their personal information will be kept completely confidential. The information records of enrolled patients will be identified with study numbers rather than names. All study members and sponsors are required to maintain confidentiality. This study will be conducted strictly in accordance with relevant Chinese regulations such as the "Ethical Review Methods for Biomedical Research Involving Humans" and international ethical guidelines such as the Declaration of Helsinki. Additionally, this study follows the tracking review of the Ethics Committee of the First Affiliated Hospital of Xi'an Jiaotong University.

ELIGIBILITY:
Inclusion Criteria:

* Meet the criteria for a family cluster of unfavorable prognoses associated with HBV infection: that is, patients with HBV infection in two consecutive generations of blood relatives, and at least one patient with cirrhosis or HCC in two or more generations of blood relatives;
* Chronic HBV-infected individuals from families with unfavorable prognoses clustering (meeting either (1)+(2) or (1)+(3) criteria): (1) Positive for HBsAg for more than 6 months; (2) Treated with nucleos(t)ide analogs (NAs); (3) Compensated cirrhosis due to hepatitis B (for details, see the "Guidelines for the Prevention and Treatment of Chronic Hepatitis B (2022 Edition)");
* A negative pregnancy test within 24 hours before the first administration of medication in the treatment group (for women of childbearing age);
* No contraindications for interferon treatment.

Exclusion Criteria:

* Patients diagnosed with liver cancer or other systemic tumors before treatment;
* Patients with contraindications to Peg IFN α-2b use (for details, see the "Guidelines for the Prevention and Treatment of Chronic Hepatitis B (2022 Edition)");
* Peripheral blood counts: WBC < 3.0 × 10^9/L, PLT < 70 × 10^9/L;
* Liver function: ALT > 5 × upper limit of normal (ULN), TBIL > 2 × ULN; Individuals planning to receive organ transplantation or who have already undergone organ transplantation;
* Those allergic to interferon or with any contraindication listed in the product information;
* Any other conditions deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted across multiple centers in China, planning to enroll 600 non-cirrhosis and 300 compensated cirrhosis patients with a family history of unfavorable prognoses clustering of HBV infection who also have HBsAg positivity for more than 6 months, and who meet the inclusion criteria and do not meet the exclusion criteria. In the non-cirrhosis cohort, the Peg IFN α-2b combination therapy group plans to enroll 300 patients, and the nucleos(t)ide group plans to enroll 300 patients; in the compensated cirrhosis cohort, the Peg IFN α-2b combination therapy group plans to enroll 150 patients, and the nucleos(t)ide group plans to enroll 150 patients.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2032-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
the number and percentage of cases of cirrhosis and HCC occurring in the non-cirrhosis population | From enrollment to the end of treatment at 5 years and 7 years
the number and percentage of cases of decompensated cirrhosis and HCC occurring in the compensated cirrhosis population | From enrollment to the end of treatment at 5 years and 7 years

SECONDARY OUTCOMES:
Overall survival time of patients in each treatment subgroup | From enrollment to the end of treatment at 5 years and 7 years
the time of cirrhosis and HCC occurring in the non-cirrhosis population | From enrollment to the end of treatment at 5 years and 7 years
the time of decompensated cirrhosis and HCC occurring in the compensated-cirrhosis population | From enrollment to the end of treatment at 5 years and 7 years
the number and percentage of HBsAg seroconversion cases, the number and percentage of HBeAg seroconversion cases (for those who are HBeAg-positive) per 24 weeks | From enrollment to the end of treatment at 5 years and 7 years
HBV DNA levels, HBsAg levels, and HBeAg levels per 24 weeks | From enrollment to the end of treatment at 5 years and 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Yingren Zhao, Professor, Study Director — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided